CLINICAL TRIAL: NCT02456844
Title: Effects of BMS-986142 on the Single-dose Pharmacokinetics of Methotrexate and Probe Substrates Montelukast (CYP2C8), Flurbiprofen (CYP2C9), Midazolam (CYP3A4), Digoxin (P-gp), and Pravastatin (OATP1B1) in Healthy Subjects
Brief Title: Study to Investigate the Effect of BMS-986142 on the Pharmacokinetics (PK) of Methotrexate and Probe Substrate Cocktail in Healthy Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IM006-003
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — montelukast; Flurbiprofen; Midazolam; Digoxin; Pravastatin; Methotrexate; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Montelukast, Flurbiprofen, Midazolam, Digoxin, Pravastatin and BMS-986142
  Interventions: Drug: Montelukast, Flurbiprofen, Midazolam, Digoxin, Pravastatin and BMS-986142
- Group 2 (Experimental): Methotrexate,Leucovorin and BMS-986142
  Interventions: Drug: Methotrexate, Leucovorin and BMS-986142

INTERVENTIONS:
Drug: Montelukast, Flurbiprofen, Midazolam, Digoxin, Pravastatin and BMS-986142 — 1. Montelukast 10-mg tablet: On Days 1 and 8,Single oral dose
  2. Flurbiprofen 50-mg tablet: On Days 1 and 8,Single oral dose
  3. Midazolam syrup 2.5 mL × 2 mg/mL (5 mg): On Days 1 and 8,Single oral dose
  4. Digoxin (Lanoxin®) 0.25 mg tablet: On Days 1 and 8,Single oral dose
  5. Pravastatin 40-mg tablet: On Days 1 and 8,Single oral dose
  6. BMS-986142: On Days 6 through 12.
  Arms: Group 1
Drug: Methotrexate, Leucovorin and BMS-986142 — 1. Methotrexate (MTX) single oral dose of 3 × 2.5-mg tablet (Days 1 and 8)
  2. Leucovorin single oral dose of 15-mg tablet (Days 2 and 9; 24 hours after MTX administration)
  3. BMS-986142 on Days 6 through 10.
  Arms: Group 2

SUMMARY:
To study the Pharmacokinetics (PK) parameters of montelukast, flurbiprofen, midazolam, digoxin, pravastatin, and MTX when coadministered with BMS-986142.

ELIGIBILITY:
Inclusion Criteria:

Groups 1 and 2:

1. Written informed consent from all subjects.
2. Body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive
3. Non-smokers.
4. Normal renal function at screening as evidenced by an estimated glomerular filtration rate (GFR) of > 90 mL/min/1.73 m2 .
5. Subject reenrollment.
6. Males who are sexually active with women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of BMS-986142.
7. Male subjects must be willing to refrain from sperm donation during the entire study plus 5 half-lives of BMS-986142.

Group 1 only:

1. Healthy male and female (not of childbearing potential) subjects as determined by medical history, and clinical assessments.
2. Women must have documented proof that they are not of childbearing potential and must not be breast feeding.

Group 2 only:

1. Healthy male subjects as determined by medical history, and clinical assessments.

Exclusion Criteria:

1. Administration of live vaccine including polio vaccine during the course of the study, 12 weeks prior to the first dose of study drug, or 30 days after the last dose of study drug.
2. Active tuberculosis (TB) requiring treatment within the previous 3 years.
3. History of herpes zoster.
4. Subjects who have experienced recent infection, upper respiratory infection,.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Days 1 through 10
Area under the plasma concentration-time curve from time zero to the time of last quantifiable concentration, AUC(0-T) | Days 1 through 10
Area under the plasma concentration-time curve from time zero extrapolated to infinite time, AUC(INF) | Days 1 through 10

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) | Days 1 through 10
Terminal plasma half-life (T-half) | Days 1 through 10
Apparent total body clearance (parents only), CLT/F | Days 1 through 10
Ratio of metabolite Cmax to parent Cmax, corrected for molecular weight | Days 1 through 10
Ratio of metabolite AUC(0-T) to parent AUC(0-T), corrected for molecular weight | Days 1 through 10
Ratio of metabolite AUC(INF) to parent AUC(INF), corrected for molecular weight | Days 1 through 10
Trough observed plasma concentration (For BMS-986142 only) | Days 1 through 10

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Hunt, MD PhD, Principal Investigator — PPD Development, LP